CLINICAL TRIAL: NCT00772928
Title: Immunogenicity Assessment of Pentacel™ (Hybrid CP20/20/5/3DT-mIPV//PRP-T) When Given at Different Times From or Concurrently With a Pneumococcal Conjugate Vaccine
Brief Title: Study of the Effect of Pneumococcal Conjugate Vaccine (PCV) on Immunogenicity of Pentacel™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M5A07
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Results first posted 2010-02-12 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Diphtheria; Tetanus; Haemophilus Infection; Pertussis; Polio
Keywords: Pertussis; Whooping cough; Diphtheria; Tetanus; Haemophilus influenzae; Poliovirus Types 1, 2, and 3.
MeSH Terms: conditions — Diphtheria; Tetanus; Haemophilus Infections; Whooping Cough; Poliomyelitis | interventions — Heptavalent Pneumococcal Conjugate Vaccine; pentacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pentacel™ concurrently with Prevnar® (Experimental): Participants had Pentacel™ concurrently administered with Prevnar®
  Interventions: Biological: Pentacel™: HCPDT-IPV//PRP-T Vaccine and Prevnar®
- Pentacel™ staggered schedule with Prevnar® (Experimental): Participants had Pentacel™ given at different times from Prevnar® (using a standardized, staggered schedule).
  Interventions: Biological: Pentacel™: HCPDT-IPV//PRP-T Vaccine and Prevnar®

INTERVENTIONS:
Biological: Pentacel™: HCPDT-IPV//PRP-T Vaccine and Prevnar® — 0.5 mL, Intramuscular
  Other Names: Pentacel™; Prevnar®
  Arms: Pentacel™ concurrently with Prevnar®
Biological: Pentacel™: HCPDT-IPV//PRP-T Vaccine and Prevnar® — 0.5 mL, Intramuscular
  Other Names: Pentacel™; Prevnar®
  Arms: Pentacel™ staggered schedule with Prevnar®

SUMMARY:
This study is designed to evaluate in a controlled manner the effect of Prevnar® on the immune responses of Pentacel™

Primary Objective - Stage I:

To compare the immune responses elicited by an infant series of Pentacel™ when given at different times from or concurrently with a Pneumococcal conjugate vaccine (Prevnar®).

Primary Objective - Stage II:

To compare the immune responses elicited by a 4th dose of Pentacel™ when given at different times from or concurrently with Prevnar®.

DETAILED DESCRIPTION:
This is a 2-staged study. Stage I of this study is designed to compare the immune responses elicited by an infant series (3 doses) of Pentacel™ when given at different times from or concurrently with Prevnar®.

Stage II is designed to describe the immune responses elicited by a 4th dose of Pentacel™ (all antigens) when given at different times from or concurrently with Prevnar®.

ELIGIBILITY:
Inclusion Criteria :

* Healthy infants 2 months (≥ 42 days and ≤ 89 days) of age.
* Infants with at least 36 weeks of gestation at delivery.
* Must have received 1 dose of Hepatitis B vaccine (with that dose at least 15 days before the administration of study vaccines).
* Able to attend the scheduled visits and to comply with the study procedures.
* Parent or legal guardian willing to take rectal temperatures during the infant series.
* Parent or legal guardian has access to a telephone.
* Signed informed consent from parent or legal guardian obtained before the 1st study intervention.
* Able to obtain at least 1.5 mL of blood sample prior to Dose 1.

Exclusion Criteria :

* Clinically significant findings on review of systems (determined by investigator or sub-investigator to be sufficient for exclusion).
* Known or suspected hypersensitivity to any component of the study vaccine to be administered.
* Known or suspected impairment of immunologic function or receipt of immunosuppressive therapy or immunoglobulin since birth.
* Known Human Immunodeficiency Virus (HIV)-positive mother or child.
* Personal or immediate family history of congenital immune deficiency.
* Developmental delay or neurologic disorder.
* Chronic medical, congenital, or developmental disease.
* Participation in any other clinical trial.
* Any condition which, in the opinion of the investigator, would interfere with the evaluation of the vaccine or pose a health risk to the subject.
* Prior history of having received any Acellular Pertussis- (DTaP) or Whole Cell Pertussis- (DTwP) based combination vaccines, Haemophilus influenzae Type b (Hib)-conjugate, Poliovirus, or Pneumococcal conjugate vaccines.

Ages: 42 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1167 (Actual)
Dates: Start 2003-10; Primary Completion 2006-05 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (22):
- United States (22):
  - Montgomery, Alabama
  - Fayetteville, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Fountain Valley, California
  - Oakland, California
  - Rolling Hills Estate, California
  - Norwich, Connecticut
  - Bardstown, Kentucky
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Kansas City, Missouri
  - Brooklyn, New York
  - Norristown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Austin, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - Layton, Utah
  - Spokane, Washington
  - Vancouver, Washington
  - La Crosse, Wisconsin

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 30 October 2003 to 29 March 2004 in 23 medical clinics in the US.
Pre-assignment Details: A total of 1167 subjects that met the inclusion and exclusion criteria were enrolled, 1166 were vaccinated.
Groups:
- Pentacel™ Concurrently With Prevnar®: Participants receieved Pentacel™ vaccine concurrently with Prevnar® vaccine
- Pentacel™ Staggered Schedule With Prevnar®: Participants received Pentacel™ vaccine at different times from Prevnar® vaccine (using a standardized, staggered schedule).
Period: Overall Study
Arm/Group | Pentacel™ Concurrently With Prevnar® | Pentacel™ Staggered Schedule With Prevnar®
Started | 587 | 579
Completed | 543 | 538
Not Completed | 44 | 41
Not completed — Lost to Follow-up | 9 | 6
Not completed — Protocol Violation | 10 | 12
Not completed — Withdrawal by Subject | 25 | 22
Not completed — Did not receive vaccine | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pentacel™ Concurrently With Prevnar® | Pentacel™ Staggered Schedule With Prevnar® | Total
Number analyzed (Participants) | 587 | 579 | 1166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 587 | 579 | 1166
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Months] | 2.2 (0.29) | 2.1 (0.28) | 2.1 (0.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 278 | 259 | 537
  Male | 309 | 320 | 629
Region of Enrollment [Number; unit: participants]
  United States | 587 | 579 | 1166

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 4-fold Rises in Levels of Pentacel™ Vaccine Antibody Titers Post-dose 3 When Given at Different Times or Concurrently With a Pneumococcal Conjugate Vaccine (Prevnar®)
Description: Seroconversion was defined as the percentage of subjects with ≥ 4-fold post-dose 3 for anti-pertussis and ≥ 0.15 μg/mL or ≥ 1.0 μg/mL for anti-Polyribosylribitol Phosphate (PRP) responses.
Time Frame: 28 to 48 days post-3rd vaccination
Population: Analysis was on the total number of subjects with available serology data from the per-protocol immunogenicity population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pentacel™ Concurrently With Prevnar® | Pentacel™ Staggered Schedule With Prevnar®
Number analyzed (Participants) | 447 | 438
Percentage of Participants
  Pertussis Toxoid (PT) EU/mL | 90 | 90
  Filamentous Haemagglutinin (FHA) EU/mL | 82 | 82
  Fimbriae Types 2 and 3 (FIM 2&3) EU/mL | 88 | 88
  Pertactin (PRN) EU/mL | 74 | 72
  Poliovirus Polyribosyl. P Tetanus, PRP ≥0.15 μg/mL | 96 | 95
  Poliovirus Polyribosyl. P Tetanus, PRP ≥0.10 μg/mL | 77 | 80

2. Primary Outcome: Geometric Mean Titers of Antibodies to Pertussis, Diphtheria, Tetanus, Polyribosylribitol Phosphate and Poliovirus Elicited by an Infant Series of Pentacel™ When Given at Different Times or Concurrently With a Pneumococcal Conjugate Vaccine (Prevnar®)
Description: Anti-pertussis response include antibodies to Pertussis Toxoid (PT); Filamentous Haemagglutinin (FHA); Fimbriae Types 2 and 3 (FIM) and Pertactin (PRN) antigens.
Time Frame: 60 Days Post-dose 3
Population: Geometric mean titer analysis was on the total number of subjects with available serology data from the per-protocol immunogenicity population
Measure: Geometric Mean (95% Confidence Interval); unit: All Units
Arm/Group | Pentacel™ Concurrently With Prevnar® | Pentacel™ Staggered Schedule With Prevnar®
Number analyzed (Participants) | 447 | 439
All Units
  Pertussis Toxoid (PT) EU/mL | 103.58 [97.87 to 109.63] | 102.78 [96.86 to 109.06]
  Filamentous Haemagglutinin (FHA) EU/mL | 82.41 [77.40 to 87.75] | 77.80 [72.62 to 83.35]
  Fimbriae Types 2 and 3 (FIM) EU/mL | 272.47 [251.39 to 295.32] | 280.97 [258.02 to 305.97]
  Pertactin (PRN) EU/mL | 45.7 [41.59 to 50.23] | 44.28 [40.11 to 48.89]
  Poliovirus Polyribosylribitol P Tetanus(PRP) μg/mL | 3.32 [2.85 to 3.87] | 3.60 [3.09 to 4.20]
  Diphtheria (IU/mL) | 0.59 [0.53 to 0.64] | 1.32 [1.22 to 1.42]
  Tetanus (IU/mL) | 1.27 [1.18 to 1.35] | 1.30 [1.21 to 1.39]
  Polio 1 (1/dil) | 543.52 [480.61 to 614.67] | 593.09 [515.54 to 682.31]
  Polio 2 (1/dil) | 846.36 [752.37 to 952.08] | 949.06 [847.95 to 1062.22]
  Polio 3 (1/dil) | 1025.73 [899.05 to 1170.26] | 1104.05 [969.80 to 1256.88]

3. Other Pre Specified Outcome: Percentage of Subjects With Solicited Local, Systemic Reactions Occurring Between 0-3 Days After Each Dose of Pentacel™
Description: Solicited local reactions: redness, swelling, and tenderness. Solicited systemic reactions: fever (temperature), irritability post-vaccinal, crying, lethargy, appetite decreased, vomiting, diarrhea, and rash.
Time Frame: 0-3 days post- vaccination and entire study period
Population: Analysis was on all enrolled and vaccinated subjects, intend-to-treat population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pentacel™ Concurrently With Prevnar® | Pentacel™ Staggered Schedule With Prevnar®
Number analyzed (Participants) | 587 | 579
Percentage of Participants
  Any Solicited Local Reaction Post-dose 1 | 31 | 26
  Any Redness Post-dose 1 | 5 | 3
  Grade 3 Redness, > 50 mm Post-dose 1 | 0 | 0
  Any Swelling Post-Dose 1 | 4 | 4
  Grade 3 Swelling, > 50 mm Post-dose 1 | 0 | 0
  Any Tenderness Post-dose 1 | 28 | 24
  Grd 3 Tenderness Cries when limb is moved Post-d 1 | 1 | 1
  Any Solicited Local Reaction Post-dose 2 | 24 | 15
  Any Redness Post-dose 2 | 4 | 4
  Grade 3 Redness, > 50 mm Post-dose 2 | 0 | 0
  Any Swelling Post-Dose 2 | 2 | 2
  Grade 3 Swelling, > 50 mm Post-dose 2 | 0 | 0
  Any Tenderness Post-dose 2 | 22 | 12
  Grd 3 Tenderness Cries when limb is moved Post-d 2 | 1 | 0
  Any Solicited Local Reaction, Post-dose 3 | 20 | 9
  Any Redness Post-dose 3 | 6 | 3
  Grade 3 Redness, > 50 mm Post-dose 3 | 0 | 0
  Any Swelling Post-Dose 3 | 2 | 2
  Grade 3 Swelling, > 50 mm Post-dose 3 | 0 | 0
  Any Tenderness Post-dose 3 | 17 | 7
  Grd 3 Tenderness Cries when limb is moved Post-d 3 | 1 | 0
  Any Solicited Local Reaction All doses | 46 | 38
  Any Redness All doses | 12 | 8
  Grade 3 Redness, > 50 mm All doses | 0 | 1
  Any Swelling All doses | 7 | 7
  Grade 3 Swelling, > 50 mm All doses | 0 | 0
  Any Tenderness All doses | 41 | 33
  Grd3 Tenderness Cries when limb is moved All doses | 2 | 1
  Any Solicited Systemic Reaction Post-dose 1 | 69 | 64
  Any Fever Post-dose 1 | 8 | 11
  Grade 3 Fever > 39.5°C Post-dose 1 | 0 | 0
  Any Lethargy Post-dose 1 | 33 | 28
  Grd3 Lethargy not interested in usual day activity | 1 | 0
  Any Vomiting Post-dose 1 | 9 | 8
  Grade 3 Vomiting, ≥ 3 episodes Post-dose 1 | 0 | 1
  Any Diarrhea Post-dose 1 | 11 | 9
  Grade 3 Diarrhea, > 5 stools Post-dose 1 | 1 | 0
  Any Crying Post-dose 1 | 31 | 29
  Grade 3 Crying, > 3 hours Post-dose 1 | 1 | 0
  Any Irritability Post-dose 1 | 53 | 52
  Grade 3 Irritability, >3 hours Post-dose 1 | 3 | 1
  Any Appetite Decreased Post-dose 1 | 18 | 11
  Grd 3 Appetite Decreased, Refuses ≥3 feeds Post-d1 | 1 | 0
  Any Solicited Systemic Reaction, Post-dose 2 | 63 | 45
  Any Fever Post-dose 2 | 19 | 16
  Grade 3 Fever > 39.5°C Post-dose 2 | 1 | 0
  Any Lethargy Post-dose 2 | 21 | 11
  Grd3 Lethargy not interested in usual day activity | 1 | 0
  Any Vomiting Post-dose 2 | 9 | 3
  Grade 3 Vomiting, ≥ 3 episodes Post-dose 2 | 1 | 0
  Any Diarrhea Post-dose 2 | 9 | 7
  Grade 3 Diarrhea, > 5 stools Post-dose 2 | 0 | 0
  Any Crying Post-dose 2 | 25 | 14
  Grade 3 Crying, > 3 hours Post-dose 2 | 1 | 1
  Any Irritability Post-dose 2 | 47 | 34
  Grade 3 Irritability, > 3 hours Post-dose 2 | 4 | 1
  Any Appetite Decreased Post-dose 2 | 15 | 8
  Grd 3 Appetite Decreased, Refuses ≥3 feeds Post-D2 | 0 | 0
  Any Solicited Systemic Reaction, Post-dose 3 | 54 | 34
  Any Fever Post-dose 3 | 20 | 16
  Grade 3 Fever > 39.5°C Post-dose 3 | 0 | 0
  Any Lethargy Post-dose 3 | 18 | 8
  Grd3 Lethargy not interested in usual day activity | 1 | 0
  Any Vomiting Post-dose 3 | 4 | 5
  Grade 3 Vomiting, ≥ 3 episodes Post-dose 3 | 0 | 0
  Any Diarrhea Post-dose 3 | 6 | 4
  Grade 3 Diarrhea, > 5 stools Post-dose 3 | 0 | 0
  Any Crying Post-dose 3 | 18 | 9
  Grade 3 Crying, > 3 hours Post-dose 3 | 0 | 0
  Any Irritability Post-dose 3 | 40 | 26
  Grade 3 Irritability, > 3 hours Post-dose 3 | 2 | 2
  Any Appetite Decreased Post-dose 3 | 11 | 7
  Grd 3 Appetite Decreased, Refuses ≥3 feeds Post-D3 | 1 | 0
  Any Solicited Systemic Reaction, All doses | 87 | 78
  Any Fever All doses | 35 | 32
  Grade 3 Fever > 39.5°C, All doses | 1 | 1
  Any Lethargy All doses | 46 | 36
  Grd3 Lethargy not interested in usual day activity | 2 | 1
  Any Vomiting All doses | 18 | 14
  Grade 3 Vomiting, ≥ 3 episodes All doses | 1 | 1
  Any Diarrhea All doses | 21 | 18
  Grade 3 Diarrhea, > 5 stools All doses | 1 | 1
  Any Crying All doses | 48 | 39
  Grade 3 Crying, > 3 hours All doses | 1 | 1
  Any Irritability All doses | 74 | 68
  Grade 3 Irritability, > 3 hours All doses | 7 | 4
  Any Appetite Decreased All doses | 33 | 21
  Grd 3 Appetite Decreased, Refuses ≥ 3 feeds All D | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from day of enrollment over a period of 5 months post-vaccination 1
Arm/Group | Pentacel™ Concurrently With Prevnar® | Pentacel™ Staggered Schedule With Prevnar®
Serious Adverse Events (participants affected / at risk) | 32/587 | 15/579
Other Adverse Events (participants affected / at risk) | 475/587 | 481/579
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentacel™ Concurrently With Prevnar® (N=587) | Pentacel™ Staggered Schedule With Prevnar® (N=579)
Lymphadenitis nos (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastrointestinal malformation nos (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Lymphangioma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Acquired pyloric stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea nos (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcers (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction nos (Gastrointestinal disorders) | 1 (1) | 0 (0)
Developmental delay nos (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 11 (11) | 10 (10)
Candidal infection nos (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Otitis media nos (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia nos (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis nos (Infections and infestations) | 1 (1) | 1 (1)
Respiratory syncytial virus infection nos (Infections and infestations) | 1 (1) | 1 (1)
Roseola (Infections and infestations) | 1 (1) | 0 (0)
Skin and subcutaneous tissue abscess nos (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection viral nos (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection nos (Infections and infestations) | 3 (3) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture nos (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Convulsions nos (Nervous system disorders) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1)
Febrile convulsion (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vesico-ureteric reflux (Renal and urinary disorders) | 1 (1) | 0 (0)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentacel™ Concurrently With Prevnar® (N=587) | Pentacel™ Staggered Schedule With Prevnar® (N=579)
Conjunctivitis (Eye disorders) | 60 (65) | 59 (67)
Constipation (Gastrointestinal disorders) | 30 (34) | 35 (40)
Diarrhoea NOS (Gastrointestinal disorders) | 28 (28) | 41 (43)
Flatulence (Gastrointestinal disorders) | 42 (51) | 41 (48)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 34 (34) | 35 (35)
Teething (Gastrointestinal disorders) | 91 (104) | 127 (154)
Pyrexia (General disorders) | 45 (55) | 29 (35)
Bronchiolitis (Infections and infestations) | 66 (70) | 75 (86)
Candidal infection NOS (Infections and infestations) | 36 (41) | 39 (43)
Gastroenteritis NOS (Infections and infestations) | 35 (40) | 41 (44)
Nasopharyngitis (Infections and infestations) | 41 (43) | 47 (55)
Otitis media NOS (Infections and infestations) | 162 (226) | 162 (244)
Otitis media serous acute NOS (Infections and infestations) | 37 (44) | 26 (33)
Upper respiratory tract infection NOS (Infections and infestations) | 258 (352) | 264 (368)
Upper respiratory tract infection viral NOS (Infections and infestations) | 24 (29) | 35 (35)
Viral infection NOS (Infections and infestations) | 46 (50) | 50 (55)
Cough (Respiratory, thoracic and mediastinal disorders) | 52 (56) | 64 (75)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 48 (50) | 55 (65)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 22 (24) | 29 (35)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 34 (39)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 23 (25) | 30 (31)
Eczema (Skin and subcutaneous tissue disorders) | 41 (41) | 33 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.